CLINICAL TRIAL: NCT04713618
Title: Longitudinal Changes in Women's Pelvic Health and Sexual Function After Pelvic Radiation
Brief Title: Changes in Pelvic Health, Sexual Function, and Quality of Life in Women With Pelvic Cancer Undergoing Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Arthur, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-19342; NCI-2020-04790 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-12-18; First posted 2021-01-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Anal Carcinoma; Cervical Carcinoma; Endometrial Carcinoma; Malignant Pelvic Neoplasm; Rectal Carcinoma; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Anus Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Pelvic Neoplasms; Rectal Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal Microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive Care (pelvic exam, survey): Patients undergo standard of care pelvic exam at baseline and 1, 3, 6, 12, and 24 month follow ups. Patients also complete patient reported outcome measures at baseline and 1, 3, 6, 12, 18, and 12 month follow ups.
  Interventions: Procedure: Pelvic Examination; Other: Survey

INTERVENTIONS:
Procedure: Pelvic Examination — Undergo pelvic exam
  Other Names: internal examination; Pelvic Exam
Other: Survey — Complete surveys
  Other Names: Survey Instrument

SUMMARY:
This study investigates changes in physical measures of pelvic health and patient-reported outcomes of sexual function, intimate relationship, and quality of life over time in women undergoing radiation therapy for pelvic cancer. Evaluating vaginal changes prior to and after a course of radiation and collecting patient reported outcomes of sexual function, partner communication, and intimacy may help researchers may help researchers better understand physical changes and symptoms over time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate changes in objective physical exam findings from baseline to the end of radiation and through two years follow-up for women with pelvic cancer.

II. To examine changes in sexual, relational and quality of life outcomes from baseline to the end of radiation and through one year follow-up for women with pelvic cancer using the patient reported outcome measures.

III. To compare physical exam and patient-reported outcome trajectories over time.

OUTLINE:

Patients undergo standard of care pelvic exam at baseline and 1, 3, 6, 12, and 24 month follow ups. Patients also complete patient reported outcome measures at baseline and 1, 3, 6, 12, 18, and 12 month follow ups.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with anal, rectal, cervical, endometrial, vaginal, or vulvar cancer receiving external beam radiation alone, brachytherapy alone, or both external beam radiation and brachytherapy
* Concurrent or prior chemotherapy is allowed, including those participating in Ohio State University (OSU)-16166
* Any prior gynecologic surgery is permitted
* Rectal surgery, including lower anterior resection and abdominoperineal resection, is permitted

Exclusion Criteria:

* Patients with scleroderma, mixed connective tissue disorder, and lupus will be excluded
* Patients who have received prior pelvic radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with gynecologic and colorectal cancers who are receiving either external beam radiation or brachytherapy from The Ohio State University James Cancer Hospital Radiation Oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical exam findings | Baseline up to 2 years after radiation therapy (RT)
  Vaginal Health Assessment (VHA) tool; vaginal length and diameter will be reported as categorical variables (Eaton et al., 2017). Estimates will be <2.5, 2.5, 3.0, 3.5, 4.0 or >4 cm. Vaginal length will be estimated based on manual exam. Estimates will be <4cm, 4-6cm, and >6cm. We will first test bivariate correlations between physical exam outcomes and categorical sociodemographic factors using Fisher's exact test at each time point. The study team will test bivariate correlations between physical exam outcomes and continuous sociodemographic factors using ANOVA at each time point. Next, the study team will employ one-tailed Wilcoxon signed-rank test to assess the effects of radiation by comparing 1-month, 3-month, 6-month, 12-month and 24-month physical exam outcomes to baseline.
Change in vulvovaginal symptoms | Baseline up to 2 year after RT
  The Vaginal Assessment Scale (VAS) and Vulvar Assessment Scale (VuAS) are tools to identify vulvovaginal symptoms over the past 4 weeks including vaginal dryness, soreness, irritation, and dyspareunia. Items are scored 0 (none) to 3 (severe) and a composite score is calculated by taking the mean of the items. Will first test bivariate correlations between patient reported outcomes and categorical sociodemographic factors using ANOVA. Will then test bivariate correlations between patient-reported outcomes and continuous sociodemographic factors using Pearson's correlation. Will employ one-tailed paired sample t-test to assess the effects of radiation by comparing patient-reported outcomes at each time point to baseline. Will also report 95% confidence intervals and effect sizes. Will utilize mixed-effects modeling to demonstrate changes in each outcome variable over time adjusting for demographic/clinical characteristics.
Change in sexual function | Baseline up to 2 year after RT
  Female Sexual Functioning Index (FSFI) is a 19 item self -reported instrument measuring six domains of sexual functioning including arousal, orgasm, satisfaction and pain. The maximum score is 36 and a score of ≤ 26.0 indicates sexual dysfunction. Will first test bivariate correlations between patient reported outcomes and categorical sociodemographic factors using ANOVA. Will then test bivariate correlations between patient-reported outcomes and continuous sociodemographic factors using Pearson's correlation. Will employ one-tailed paired sample t-test to assess the effects of radiation by comparing patient-reported outcomes at each time point to baseline. Will also report 95% confidence intervals and effect sizes. Will utilize mixed-effects modeling to demonstrate changes in each outcome variable over time adjusting for demographic/clinical characteristics.

SECONDARY OUTCOMES:
Change in vaginal microbiome | Baseline up to 2 year after RT
  The Lactobacillus to Prevotella ratio (LPR) will be calculated. The vaginal dryness (binary, VAS score <=2 vs >2) will be related to the LPR (continuous) by logistic regression. A significant relationship of LPR with vaginal dryness will be evaluated by Wald test. The LPR is correlated with abundance of macrophages by Spearman correlation. Spearman correlation is used to determine the association between LPR relative abundance and expression of a gene or composition of the immune cells. We will use linear discriminant analysis to explore a linear combination of gene expression, microbe relative abundance and immune cell composition to predict vaginal dryness. The level of inflammation in the tissue will be estimated by aggregating the expression of standard "inflammasome" genes. LPR will be correlated with the aggregated inflammation value by Spearman correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Arthur, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu